CLINICAL TRIAL: NCT00575484
Title: Hypertonic Saline With Furosemide and a Normosodic Diet for the Treatment of Decompensated Congestive Heart Failure With Prerenal Physiology
Brief Title: Concentrated Saline Infusions and Increased Dietary Sodium With Diuretics for Heart Failure With Kidney Dysfunction
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Barnes-Jewish Hospital (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Anitha Vijayan, MD, Professor of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00904-0407-01
Record Dates: First submitted 2007-12-17; First posted 2007-12-18 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Congestive Heart Failure; Renal Insufficiency
Keywords: Congestive Heart Failure; Renal Insufficiency; Hypertonic Saline Solution; Diuretic Resistance; Cardiorenal Syndrome
MeSH Terms: conditions — Heart Failure; Renal Insufficiency; Cardio-Renal Syndrome | interventions — Saline Solution, Hypertonic; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Normal saline, then oral placebo capsule
- 2 (Active Comparator)
  Interventions: Drug: Hypertonic saline, then oral sodium chloride

INTERVENTIONS:
Drug: Hypertonic saline, then oral sodium chloride — 2mL/kg hypertonic saline (4.4% NaCl if serum sodium </=135, else 2.8% NaCl) infused over 30min BID and dosed simultaneously with IV bolus furosemide BID (latter dose per treating physician) until patient is switched to oral loop diuretic. After switch to oral diuretic, subject will receive oral 0.75gm sodium (NaCL) capsule dosed BID with loop diuretic (latter dose per treating physician) until 60d after discharge.
  Arms: 2
Drug: Normal saline, then oral placebo capsule — 20mL normal saline infusion X 30min BID dosed simultaneously with IV bolus furosemide BID (latter dose per treating physician) PLUS 2gm sodium diet PLUS 1.5L fluid restriction. After switch to oral diuretic, begin oral placebo capsule BID, dosed with loop diuretic (dose per treating physician) PLUS 2gm sodium diet PLUS 1.5L fluid restriction.
  Arms: 1

SUMMARY:
At present the standard management of fluid overload in patients with congestive heart failure (CHF) involves limiting the intake of salt and water while administering high dose diuretics, often at the cost of deteriorating kidney function. However, another group of researchers has previously shown that intravenously infusing small volumes of concentrated saline during diuretic dosing and liberalizing dietary salt intake while continuing to limit water consumption resulted in improved fluid removal in CHF patients. Furthermore, less deterioration in kidney function, shorter hospitalizations, reduced readmission rates, and even reduced mortality were observed. The present study will examine this novel therapy in a population of 60 patients with underlying severe CHF and kidney dysfunction hospitalized for the management of fluid overload. Half of these patients will receive investigational treatment with concentrated salt infusions and liberalized salt consumption during diuretic therapy. All patients will otherwise receive the standard therapies for heart failure, including restrictions on water consumption. This study will attempt to verify the improvements in clinical endpoints previously described and define the mechanisms of enhanced fluid removal.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥18) admitted with CHF exacerbation with NYHA Class III-IV symptoms at screening.
* Left ventricular ejection fraction </= 45%, as determined by previous echocardiogram, left ventricular angiogram, or thallium myocardial imaging.
* Estimated GFR <60 ml/min/1.7m² with significant prerenal physiology as judged by prior documented volume mediated changes in renal function, a fractional excretion of urea <35%, or a fractional excretion of sodium <1%. For GFR 30-60: must have serum sodium </= 135 mEq/L OR large home diuretic dose (total daily loop diuretic dose >/= 120 mg/d in furosemide equivalents OR concomitant thiazide use). For GFR <30: no additional criteria needed.

Exclusion Criteria:

* Admit estimated GFR < 15mL/min or predicted need for chronic hemodialysis within the next 60 days.
* Cause of acute kidney injury other than prerenal physiology.
* No loop diuretic prior to admission or loop diuretic initiated within the 2 wks prior to admission.
* Medicine or dietary noncompliance expected to prevent successful study participation.
* > 36hrs since presentation to screening.
* Serum Na > 145 mEq/L OR < 120 mEq/L at screening.
* Systolic blood pressure > 180 mmHg at screening.
* Presentation with acute coronary syndrome OR left heart catheterization planned at screening.
* Current or impending respiratory failure at screening.
* Current calcineurin inhibitor or nesiritide use.
* Nephrotic-range proteinuria.
* Clinical evidence for the presence of cirrhosis with bilirubin >/= 2mg/dL or international normalized ratio (not on coumadin) >/= 1.7.
* Presence of another active medical issue which may prolong hospital admission or delay aggressive CHF therapy.
* Participation in another interventional study.
* Pregnancy.
* Prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
duration of hospitalization | duration of hospitalization
weight loss at discharge | duration of hospitalization
weight loss at 60 days | 60 days after discharge

SECONDARY OUTCOMES:
number of readmissions | 60 days after discharge
GFR by creatinine clearance at discharge | duration of hospitalization
estimated GFR at 60 days after discharge | 60 days after discharge
24hr urine output at discharge | last 24hrs of hospitalization
need for inotrope or extracorporeal volume removal | 60 days after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Anitha Vijayan, M.D., Principal Investigator — Renal Division, Washington University School of Medicine; Kamalanathan K Sambandam, M.D., Principal Investigator — Renal Division, Washington University School of Medicine; Gregory A Ewald, M.D., Principal Investigator — Cardiovascular Division, Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital; Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Paterna S, Parrinello G, Amato P, Dominguez L, Pinto A, Maniscalchi T, Cardinale A, Licata A, Amato V, Licata G, Di Pasquale P. Tolerability and efficacy of high-dose furosemide and small-volume hypertonic saline solution in refractory congestive heart failure. Adv Ther. 1999 Sep-Oct;16(5):219-28. PMID 10915397
- [Background] Paterna S, Di Pasquale P, Parrinello G, Amato P, Cardinale A, Follone G, Giubilato A, Licata G. Effects of high-dose furosemide and small-volume hypertonic saline solution infusion in comparison with a high dose of furosemide as a bolus, in refractory congestive heart failure. Eur J Heart Fail. 2000 Sep;2(3):305-13. doi: 10.1016/s1388-9842(00)00094-5. PMID 10938493
- [Background] Licata G, Di Pasquale P, Parrinello G, Cardinale A, Scandurra A, Follone G, Argano C, Tuttolomondo A, Paterna S. Effects of high-dose furosemide and small-volume hypertonic saline solution infusion in comparison with a high dose of furosemide as bolus in refractory congestive heart failure: long-term effects. Am Heart J. 2003 Mar;145(3):459-66. doi: 10.1067/mhj.2003.166. PMID 12660669
- [Background] Paterna S, Di Pasquale P, Parrinello G, Fornaciari E, Di Gaudio F, Fasullo S, Giammanco M, Sarullo FM, Licata G. Changes in brain natriuretic peptide levels and bioelectrical impedance measurements after treatment with high-dose furosemide and hypertonic saline solution versus high-dose furosemide alone in refractory congestive heart failure: a double-blind study. J Am Coll Cardiol. 2005 Jun 21;45(12):1997-2003. doi: 10.1016/j.jacc.2005.01.059. PMID 15963399